CLINICAL TRIAL: NCT04808973
Title: A Pilot Study on the Efficacy of DTG Plus 3TC for Prophylaxis of Mother-to-child Transmission of HIV Infection in Pregnant Women Who Have Detectable Viral Load After 14 Weeks of Gestation
Brief Title: DTG Plus 3TC for Prophylaxis of Mother-to-child Transmission of HIV Infection in Pregnant Women
Acronym: PREGNANCY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundação Bahiana de Infectologia (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 213477
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: HIV Infections; Pregnancy Related; Mother to Child Transmission
Keywords: HIV; Pregnant women; MTCT
MeSH Terms: conditions — HIV Infections | interventions — dolutegravir; Lamivudine

STUDY DESIGN:
Intervention Model Description: A group of 20 pregnant women will be enrolled, in two phases: the first one will include 10 women, and if no safety sign is detected after completion of this initial group, additional 10 women will be enrolled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lamivudine plus Dolutegravir in FDC (Experimental): Single arm of 3TC+DTG for treatment of pregnant women with HIV infection
  Interventions: Drug: Dolutegravir plus lamivudine in a FDC

INTERVENTIONS:
Drug: Dolutegravir plus lamivudine in a FDC — All participants will receive an ART regimen composed by Lamivudine plus Dolutegravir in a single pill (FDC)

SUMMARY:
The study aims to evaluate the safety and efficacy of a 2 drugs ART regimen (lamivudine plus dolutegravir) for prevention of mother to child transmission in pregnant women with HIV. 20 pregnant women will be enrolled in this proof of concept protocol. They will be prescribed DTG-3TC (fixed-dose combination), and will be followed up to the end of gestation. Initially, a total of 10 pregnant women will be recruited for the first phase of the study. Once the first phase is successfully completed, 10 additional participants will be included in a second step.

DETAILED DESCRIPTION:
Main endpoints:

Primary:

-Proportion of women with undetectable HIV-1 plasma viral load at delivery

Secondary:

* Proportion of women switching therapy up to delivery
* Frequency of adverse events, regardless its relationship to the ARV drugs, for mothers and babies Frequency of MTCT

Inclusion criteria:

* Confirmed HIV infection
* No previous exposure to ARV drugs
* Plasma viral load ≥1,000 copies/ml
* Gestational age ≥ 14 and ≤ 28 weeks (checked by ultrasound)
* Age ≥ 15 years Exclusion criteria
* Presence of genotypic resistance mutations for 3TC or DTG
* Presence of active Hepatitis C
* Hepatitis B infection (a positive test for HBcore or HBsurface antibodies)
* Anemia (haemoglobin less than 8 g/dL);
* Need to use concomitant drugs with potentially relevant DDI, which require DTG dose adjustment (e.g., rifampin, carbamazepine, phenobarbital,phenytoin)
* Elevations in serum levels of alanine aminotransferase (ALT) greater than 5 times the upper limit of normal (ULN) or ALT >3xULN and bilirubin >1.5ULN (with >35% direct bilirubin);
* A history or clinical suspicion of unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hyperbilirubinaemia, oesophageal or gastric varices or persistent jaundice);
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Presence of severe pre-eclampsia, or other pregnancy related events such as renal or liver abnormalities (grade 2 or above proteinuria, elevation in serum creatinine CrCl<50 ml/min), total bilirubin, ALT or AST); After providing a written informed consent the woman will be prescribed a 2D regimen (3TC+DTG). They will be evaluated at baseline, and every 4 weeks, up to delivery.

Baseline Screening All consenting participants will have the following information and measurements collected at baseline.

* Demographics, including education.
* Documentation of HIV infection.
* CD4+ cell count and CD4%: one measurement within 60 days before inclusion.
* Targeted health history including date of first diagnosis of HIV infection, likely mode of HIV infection, history of non-AIDS events, history of sexually transmitted diseases (STIs) and gestational age.
* Brief clinical evaluation including weight, height, sitting blood pressure, pulse, and smoking status.
* Nadir CD4+ cell count and CD4% and maximum HIV RNA level available in the medical record from any time in the past.
* Findings from previous genotypic or other form of HIV resistance testing (such as virtual phenotype and/or phenotypic resistance testing), if performed and available.
* Concomitant medications, including any herbal/traditional remedies.
* Use of alcohol and recreational drugs.
* HIV transmission risk behavior assessment.
* HIV RNA measurement within the 4 previous weeks.

Additional laboratory assessments (participants should be asked to abstain from food, except water, for at least 8 hours prior to providing blood for glucose and lipid measurements):

* Complete blood count (CBC): hemoglobin, hematocrit, white blood cell count (WBC) with differential and platelets.
* CD8+ T-cell count and CD8%.
* Renal function: serum creatinine to estimate GFR.
* Liver function: alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase, total bilirubin and albumin.
* Glucose and glycosylated Hb
* Lipids: total cholesterol, low density lipoprotein (LDL), high density lipoprotein (HDL), triglycerides.
* Dipstick urinalysis for measurement of protein.
* Documentation of hepatitis B and C status: hepatitis B surface antigen, core antibody and surface antibody; hepatitis C antibody and, if available, genotype and viral load. Documented positive tests at any time in the past or documented negative tests in the 6 months before study entry may be used.
* HIV resistance testing Besides the routine medical evaluation they will be asked to provide a blood sample at every medical visit (every 4 weeks) to assess WBC, platelets count, hemoglobin, creatinine, liver enzymes, and fasting glucose / lipids. HIV-1 plasma viral load will also be assessed at the same time intervals. CD4/CD8+ cells count will be measured at baseline and after 24 and 36 weeks of gestation, or more frequently, at medical discretion.

According to the Brazilian MOH recommendations, babies will receive oral AZT for 4 weeks, if their mothers had a documented HIV RNA plasma viral load <1,000 copies/ml, in the third trimester of gestation. For those born from mothers presenting higher viral load, nevirapine will be added for the same period of time. In addition, they will be evaluated at delivery, after 2 and 6 weeks after the end of prophylaxis for HIV viral load measurements. Blood chemistry and hematology will be assessed 2 weeks after prophylaxis.16,17

Stopping criteria:

Participants will be excluded from study if the following conditions are met:

a) HIV-1 plasma viral load decay < 1 log compared with baseline values after 4 weeks of therapy, OR b) HIV-1 plasma viral load ≥ 1,000 copies/mL after 8 weeks of therapy Women will be recruited in a stepwise approach. Initially, 10 participants will be included, and followed up to the end of pregnancy. An interim analysis will evaluate the efficacy of the 2D ART regimen after the first 10 patients given birth. The study will be interrupted if 3 participants meet stopping criteria.

The second phase will start only if the number of women achieving the stopping criteria is ≤ 3 at completion of follow up for the first 10 participants, and will include 10 additional participants.

The study will have an estimated recruitment period of 4 months plus a maximum 6 months of follow up for the last enrolled patient, for each phase. Taken together, the first and second phases will require 20 months for enrollment and follow up. An interim analysis following the first phase will take one month, and the final analysis / writing reports is planned to last 3 months. Thus, the total duration of the study will be 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HIV infection
* No previous exposure to ARV drugs
* Plasma viral load ≥1,000 copies/ml
* Gestational age ≥ 14 and ≤ 28 weeks (checked by ultrasound)
* Age ≥ 15 years

Exclusion Criteria:

* Presence of genotypic resistance mutations for 3TC or DTG
* Presence of active Hepatitis C
* Hepatitis B infection (a positive test for HBcore or HBsurface antibodies)
* Anemia (haemoglobin less than 8 g/dL);
* Need to use concomitant drugs with potentially relevant DDI, which require DTG dose adjustment (e.g., rifampin, carbamazepine, phenobarbital,phenytoin)
* Elevations in serum levels of alanine aminotransferase (ALT) greater than 5 times the upper limit of normal (ULN) or ALT >3xULN and bilirubin >1.5ULN (with >35% direct bilirubin);
* A history or clinical suspicion of unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hyperbilirubinaemia, oesophageal or gastric varices or persistent jaundice);
* Subjects with severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Presence of severe pre-eclampsia, or other pregnancy related events such as renal or liver abnormalities (grade 2 or above proteinuria, elevation in serum creatinine CrCl<50 ml/min), total bilirubin, ALT or AST)

Min Age: 15 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — only pregnant women will be included
Enrollment: 20 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
undetectable HIV-1 plasma viral load at delivery | 6 months
  proportion of women achieving a plasma HIV RNA viral load below 50 copies at delivery

SECONDARY OUTCOMES:
switch fo therapy up to delivery | 6 months
  proportion of women switching therapy before delivey, any reason
frequency of adverse events for mothers and babies | 8 months
  Frequency of adverse events, regardless its relationship to the ARV drugs, for mothers and babies

CONTACTS AND LOCATIONS:
Locations (1):
- Fundação Bahiana de Infectologia, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: No